CLINICAL TRIAL: NCT05397106
Title: Post-Market Clinical Follow-up of Patients With CODMAN CERTAS Plus Programmable Valve
Brief Title: Post Market Clinical Follow-up of CODMAN CERTAS Programmable Valve
Status: Recruiting | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-CERTAS-002
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hydrocephalus; Hydrocephalus in Children; NPH (Normal Pressure Hydrocephalus); IIH - Idiopathic Intracranial Hypertension; Brain Tumor; Post-Traumatic Hydrocephalus; Hemorrhagic Stroke
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure; Pseudotumor Cerebri; Brain Neoplasms; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CODMAN CERTAS Programmable Valves: CODMAN CERTAS Plus Programmable Valve, CODMAN CERTAS Plus Small Inline Programmable Valve, and CODMAN CERTAS Plus Right Angle Programmable Valve.
  Interventions: Device: CODMAN CERTAS Plus Programmable Valve

INTERVENTIONS:
Device: CODMAN CERTAS Plus Programmable Valve — Patients will undergo implantation of the CODMAN CERTAS Plus Programmable Valve according to the device label.

SUMMARY:
Post-Market Clinical Follow-up Registry of Patients with CODMAN CERTAS Plus Programmable Valves.

DETAILED DESCRIPTION:
The CODMAN CERTAS Plus Programmable Valve is a single use implantable device designed for shunting cerebrospinal fluid (CSF) for the treatment of hydrocephalus.

The valve can be set to 8 different performance settings for intraventricular pressure and drainage of CSF. The performance setting of the valve can be set preoperatively and can also be noninvasively changed post-implantation.

This clinical investigation will maintain data for each patient from the date of implant through 3 years post-implantation.

Data collection for each patient will occur per standard of care.

However, the clinical investigation specifically aims to collect and analyze data from the day of procedure, and post-operatively at 1 month, 3 months, 6 months, 12 months, 24 months, and 36 months.

Data from follow-up visits will be analyzed according to pre-defined time-intervals referring to these follow-up moments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or legally authorized representative has agreed to participate in the study by signing the EC-approved consent form, where applicable.
2. Patients (of any age) who underwent or who plan to have a surgical procedure utilizing one of the Codman CERTAS Plus Programmable Valves.
3. Patient (legally designated representative) is willing to comply with the study protocol timelines & requirements.
4. For patients who have had the Codman CERTAS Plus Programmable Valve implanted prior to study enrollment, have available data from implantation to the current time.

Exclusion Criteria:

1. Patients undergoing implantation of the CODMAN CERTAS Plus Programmable Valve as a revision procedure.
2. Patient's planned shunt has distal drainage to the heart.
3. Patient has ventriculitis, peritonitis or meningitis.
4. Patient has sepsis.
5. Patient has a history of poor wound healing.
6. Patient has symptoms pertaining to a skin infection at or near the site of any incisions; an ear infection on either side; a respiratory tract infection; or a urinary tract infection that, in the Investigator's opinion is clinically significant and might compromise the outcome of this study.
7. Patient has had any form of bowel surgery 30 days prior to device implant or anticipates bowel surgery within 90 days following device implant.
8. Patient is otherwise determined by the Investigator to be medically unsuitable for participation in this study.
9. Patient is currently enrolled in another drug or device trial or has been previously entered in this trial.
10. Patient is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator.
11. Patients with known hypersensitivity to rifampin or clindamycin hydrochloride. This criterion applies for patients to be treated with the BACTISEAL Catheters (included in some models of the valve) only.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients of any age, gender, and ethnicity, with hydrocephalus.
  Patients will receive the CODMAN CERTAS Plus Programmable Valve type most applicable for their condition, as determined by their clinician.
Sampling Method: Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Precise Device Placement: Maintaining Integrity and Functionality at 30 Days Post-Deployment | 30 Days
  Device Success is defined as:
  1. Deployment with the correct valve positioning
  2. Original intended device in place, and
  3. No additional surgical or interventional procedures related to access or the device since completion of the original procedure.

OTHER OUTCOMES:
Incidence of Valve Replacement | 12, 24 and 36 Months
  Incidence of Valve replacement post - implantation
Adverse Events | 12, 24 and 36 Months
  Incidence of Adverse Events post - implantation
  Long term safety will be assessed by the incidence of all adverse events/complications including number of subjects with shunt and/or shunt system infections.
Number of encounters with inadvertent reprogramming of CODMAN CERTAS Plus Programmable Valves | 12, 24 and 36 Months
  Incidence of inadvertent reprogramming of CODMAN CERTAS Plus Programmable Valves post - implantation prior to MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sherese Fralin, MSN, FNP, PhD, Study Director — Integra LifeSciences
Locations (9):
- Belgium (2):
  - University Hospital Leuven, Leuven
  - AZ Delta - Roeselare, Roeselare
- Germany (5):
  - Klinikum Dortmund Wirbelsäulenchirurgie, Dortmund
  - Heinrich Heine University, Dept of Neurosurgery, Universitätsklinik Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Freiburg University Hospital, Freiburg im Breisgau
  - Katharinenhospital - Neurochirurgische Klinik Stuttgart, Stuttgart
- Hospital12 de Octubre, Madrid, Spain
- Canton Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No